CLINICAL TRIAL: NCT00376532
Title: Role of Matrix Metaloproteinase(MMP)9 and MMP 2 in Risk Stratification for Ventricular Tachycardia/Fibrillation in Patients With Implanted Cardioverter Defibrillator (ICD) Devices.
Brief Title: Extracellular Matrix Marker of Arrhythmia Risk (EMMA)
Acronym: EMMA
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: TJU 06U.282
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Myocardiopathies; Ischemia, Myocardial; Arrythmia; Death, Sudden, Cardiac
Keywords: Cardiac Ischemia; Cardiac Arrhythmia; Defibrillator; Matrix Metalloproteinase; Genetic Polymorphism
MeSH Terms: conditions — Cardiomyopathies; Myocardial Ischemia; Arrhythmias, Cardiac; Death, Sudden, Cardiac; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ICD pacing or shock event: Subjects who experienced a device treatment, defined as a pacing event or a shock event
- No ICD pacing or shock event: Subjects who did not experience a treatment defined as a pacing event or a shock event

SUMMARY:
Assess whether serum levels of MMP 2 and or MMP 9 correlate with episodes of ventricular tachycardia or fibrillation in patients who have implantable cardioverter defibrillator devices.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) is responsible for 300,000-450,000 deaths per year in the United States. While it is well known that patients with both ischemic and non-ischemic cardiomyopathy (ICM, NICM) are at increased risk for SCD, there is little beyond ejection fraction which has proven useful as a noninvasive predictor to risk stratify these patients.

Myocardial scar has been validated as an arrhythmic substrate in ischemic populations; the majority of successful ablations for lethal ventricular arrhythmias are performed on tissues in peri-infarct regions. Scar provides an anatomic electrical boundary where peri-infarct zones may lead to areas of slow conduction due to the disruption of inter-myocyte electrical conduction.

Myocardial scar is a less organized collagen deposition which disrupts the typical cardiac extracellular matrix. The collagen matrix provides mechanical support to the myocardium dictating ventricular shape, size and stiffness. While typically relatively dormant, the fibrillar collagen matrix reflects a dynamic relationship between collagen synthesis mediated by fibroblasts and collagen degradation performed by matrix metalloproteinases (MMP).

A marker for scar burden or a marker which could assess a patient's predilection to form scar after either an ischemic or non-ischemic insult may be useful in further risk stratifying this population. Since MMP levels may fluctuate in the course of ischemic or nonischemic injury a static promoter sequence which confers a higher level of MMP expression to an ischemic or nonischemic insult may prove to be a reliable marker. Functional polymorphisms of the MMP-9 gene promoters have been shown in multivariate analysis to be an independent predictor of cardiac mortality regardless of the mechanism of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* LVEF of ≤ 35% measured within 6 months of ICD implantation
* NYHA class II-IV at the time of ICD implantation
* ICD implantation at least 1 year prior to enrollment

Exclusion Criteria:

* Status post heart transplant
* Known malignancy in the past 2 years.
* Recent procedure, intervention or surgery within the past 90 days
* Acute MI, CABG, or PTCA/stent within the past 2 months.
* Active rheumatoid arthritis or pulmonary or hepatic fibrosis.
* Taking chronic steroid therapy for a medical condition
* Currently pregnant
* Enrolled in a concurrent study that may confound the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients or outpatients with the cardiac device of interest implanted prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Whellan, MD MHS FACC, Principal Investigator — Thomas Jefferson University
Locations (1):
- Jefferson Heart Institute, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with Implanted Cardiac Defibrillators were enrolled from the Heart Institute Outpatient Clinic or from the inpatient Electrophysiology Lab at Thomas Jefferson University Hospital
Groups:
- ICD Event: Subjects who experienced a device treatment, defined as a pacing event or a shock event
- No ICD Event: Subjects who did not experience a treatment defined as a pacing event or a shock event
Period: Overall Study
Arm/Group | ICD Event | No ICD Event
Started | 31 (Subjects with an event were enrolled beginning 09/14/2006.) | 32 (Subjects without an event were enrolled beginning 09/15/2006.)
Completed | 25 (Last event subject enrolled 2/22/2008) | 26 (Last non-event subject enrolled 3/18/2008.)
Not Completed | 6 | 6
Not completed — Lack sufficient blood sample | 6 | 6

BASELINE CHARACTERISTICS:
Population: Baseline analysis population was determined by the enrolled subjects for whom the MMP2 and MMP9 assays were completed.
Groups:
- Total: Total of all reporting groups
Arm/Group | ICD Pacing or Shock Event | No ICD Pacing or Shock Event | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 8 | 21
  >=65 years | 12 | 18 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: MMP-2
Description: Serum MMP-2 levels determined by Aushon Biosystems Searchlight® Protein Array Analysis.
Time Frame: At time of enrollment
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | ICD Pacing or Shock Event | No ICD Pacing or Shock Event
Number analyzed (Participants) | 25 | 26
pg/ml | 173493.4 (110996.7) | 139012.4 (68988.4)

2. Primary Outcome: MMP-9
Description: Serum MMP-9 levels determined by Aushon Biosystems Searchlight® Protein Array Analysis.
Time Frame: At time of enrollment
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | ICD Pacing or Shock Event | No ICD Pacing or Shock Event
Number analyzed (Participants) | 25 | 26
pg/ml | 1033545.8 (1351216.4) | 680388.5 (992423.6)

ADVERSE EVENTS:
Arm/Group | ICD Pacing or Shock Event | No ICD Pacing or Shock Event
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No